CLINICAL TRIAL: NCT06949020
Title: Efficacy and Safety of JMKX003142 Injection in Heart Failure Patients With Volume Overload：A Phase II, Randomized, Double-blind, Placebo-controlled Study
Brief Title: A Dose-finding Study of JMKX003142 in Treatment of Cardiac Edema
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JMKX003142-H201
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Edema
Keywords: fluid retention; heart failure
MeSH Terms: conditions — Edema, Cardiac; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- low dose group (Experimental)
  Interventions: Drug: JMKX003142 Injection
- median dose group (Experimental)
  Interventions: Drug: JMKX003142 Injection
- high dose group (Experimental)
  Interventions: Drug: JMKX003142 Injection
- placebo group (Placebo Comparator)
  Interventions: Drug: JMKX003142 placebo

INTERVENTIONS:
Drug: JMKX003142 Injection — JMKX003142 injection for experimental groups once daily for five days.
  Arms: high dose group
Drug: JMKX003142 Injection — JMKX003142 injection for experimental groups once daily for five days.
  Arms: low dose group
Drug: JMKX003142 Injection — JMKX003142 injection for experimental groups once daily for five days.
  Arms: median dose group
Drug: JMKX003142 placebo — JMKX003142 placebo for placebo groups once daily for five days.
  Arms: placebo group

SUMMARY:
To Evaluate the Safety, Efficacy, and Pharmacokinetic/Pharmacodynamics Characteristics of JMKX003142 injection Administered Randomly,Double-blind, Placebo-controlled Study in Chinese Cardiacl Edema Patients.

ELIGIBILITY:
Inclusion Criteria:

1. Can fully understand the purpose and process of the study and voluntarily sign the informed consent form;
2. Age ≥ 18 years old when signing the informed consent form;
3. At the screening stage, it has been definitely diagnosed as heart failure, and it is combined with one of the following clinical manifestations related to body fluid retention: edema of both lower limbs, jugular vein engorgement, pulmonary congestion;
4. The screening phase is currently undergoing or preparing to use one of the following diuretic therapy as background treatment during the run-in period:

1) At least 40mg/day of furosemide equivalent loop diuretics; 2) Any dose of loop diuretics combined with thiazide diuretics; 3) Any dose of loop diuretics combined with aldosterone receptor antagonists or other potassium sparing diuretics.

5. After the background treatment in the run-in period, the subject still has the following two conditions:

1. One of the following clinical manifestations related to fluid retention still exists after the induction phase treatment: edema of both lower limbs, jugular vein dilatation, pulmonary congestion;
2. During the import phase, the weight of D-1 does not change by more than 1.0 kg compared to D-3.

Exclusion Criteria:

1. Edema caused by diseases other than heart failure；
2. Subjects with ventricular assist devices during screening;
3. Subjects diagnosed with active myocarditis, myocardial amyloidosis, hypertrophic cardiomyopathy (excluding dilated phase), or valve disease with obvious valve stenosis during screening;
4. Acute myocardial infarction occurred within 30 days prior to screening; subjects with a history of persistent ventricular tachycardia or ventricular fibrillation within the 30 days prior to screening (those without implantable defibrillators); History of cerebrovascular disease within 6 months prior to screening (excluding asymptomatic cerebral infarction);
5. Subjects with hypovolemia or suspected hypovolemia;
6. Subject cannot feel thirst or have difficulty in fluid intake during screening;
7. During screening, the systolic blood pressure is less than 90mmHg or the diastolic blood pressure is less than 60mmHg;
8. Administered with tolvaptan 14days before randomization ；
9. Pregnancy (female pregnancy test positive) or lactation period;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 160 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
body weight | 5 days

IPD SHARING:
Plan to Share IPD: No